CLINICAL TRIAL: NCT04163354
Title: Glass Ionomer Sealant Versus Fluoride Varnish Application to Prevent Occlusal Caries Among Preschool Children - a Randomized Controlled Trial
Brief Title: Glass Ionomer Sealant Versus Fluoride Varnish on Occlusal Caries Prevention
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: The University of Hong Kong (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Principal Investigator, Professor Cynthia Kar-Yung Yiu, Clinical Professor in Paediatric Dentistry, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HMRF project 16172221
Record Dates: First submitted 2019-11-12; First posted 2019-11-14 (Actual); Last update posted 2019-11-14 (Actual); Status verified 2019-11

CONDITIONS: Pit and Fissure Caries; Glass Ionomer Cements; Tooth, Deciduous; Child
Keywords: Pit and Fissure Sealant; Fluorides, Topical
MeSH Terms: conditions — Van der Woude syndrome | interventions — sodium fluoride topical preparation; Fuji VII

STUDY DESIGN:
Intervention Model Description: A parallel design model with 2 treatment arms:
  1. NaF varnish: Application of a 5% NaF varnish (Duraphat, Colgate-Palmolive Ltd, Waltrop, Germany) on the occlusal surfaces of primary second molars and all other teeth, every 3 months during the study period;
  2. GI sealant: Glass ionomer sealant (GC Fuji VII® (pink)) on all primary second molars included in the studies, with no further repair/replacement of the sealant
Masking Description: Blinding is not possible as pink glass ionomer sealants will be placed on the primary molars of one of the groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NaF varnish (Active Comparator): Application of a 5% NaF varnish (Duraphat, Colgate-Palmolive Ltd, Waltrop, Germany) on the occlusal surfaces of primary second molars and all other teeth, every 3 months during the study period;
  Interventions: Procedure: 5% sodium fluoride varnish (NaF)
- GI sealant (Experimental): Glass ionomer sealant (GC Fuji VII® (pink)) on all primary second molars included in the studies, with no further repair/replacement of the sealant
  Interventions: Procedure: Glass ionomer sealant (GIS)

INTERVENTIONS:
Procedure: 5% sodium fluoride varnish (NaF) — In the NaF varnish groups, 0.25mL (one drop) of the varnish is placed in a plastic dappen dish. A disposable microbrush is used to apply the varnish onto the second primary molars included in the study and all other teeth. The child is instructed not to eat or drink after the application of varnish for at least half an hour.
  Other Names: Topical fluoride varnish; Duraphat, Colgate-Palmolive Ltd, Waltrop, Germany
  Arms: NaF varnish
Procedure: Glass ionomer sealant (GIS) — Glass ionomer sealants (GIS) is applied using the finger pressure technique described in the WHO manual for atraumatic restorative treatment (ART) (Frencken et al.; 1997). The primary second molars are cleaned by applying GC cavity conditioner with micro-applicator for 10-15 seconds, then clean with wet cotton pellets for several times. The surface will be dried with cotton pellets. GIS (GC Fuji VII) is mixed in standardized proportion with an amalgamator, then applied to the occlusal surface and slightly overfilled. A gloved finger with petroleum jelly will be used to push and rub the materials into the pits and fissures, and removing the excess. GIS will be covered and protected by a layer of petroleum jelly (Vaseline ®).
  Other Names: GC Fuji VII® (pink)
  Arms: GI sealant

SUMMARY:
The current study compares the efficacy of glass ionomer fissure sealant versus topical application of 5% sodium fluoride varnish in prevention of occlusal caries among preschool children.

DETAILED DESCRIPTION:
Topical fluoride varnish (TFV) with 5% sodium fluoride in its content has proven effective in preventing caries among children and adolescents. Its reduction in DMFT is well supported by Cochrane reviews and clinical trials. However, its effect in preventing pit and fissure caries in primary dentition has not been assessed.

Pit and fissure sealants have been a recommended procedure in preventing caries development in permanent molars. Multiple systematic reviews and clinical trials have concluded that fissure sealants are significantly more effective than topical fluoride varnishes in preventing occlusal caries in permanent molars. However, a recent Cochrane review suggested that there was still insufficient evidence to determine superiority of resin or glass ionomer fissure sealants over topical fluoride varnishes for occlusal caries prevention, due to the lack of reliable results and low quality of evidence.

Also, most studies were conducted on permanent first molars among school children, whom cooperation and moisture control can be easily achieved. However, application of fissure sealants, especially resin-based sealant, in very young children can be a technique-sensitive procedure. Compared with a mean treatment time of less than 3 minutes for varnish application, application of resin-based sealants required over 15 minutes. Moisture control is also of paramount importance for the retention and success of resin-based sealants, which may be difficult among young preschool children.

Glass-ionomer sealants can chemically bond to enamel and are more tolerable to inadequate moisture control. As its application requires less clinical steps, glass-ionomer sealant is comparatively more acceptable to younger patients and can be used in outreach settings with a large number of participants. The fluoride releasing ability is also beneficial in preventing caries especially at adjacent tooth surfaces. However, its retention rate is significantly lower than that of resin-based sealants, its success rate in preventing fissure caries in very young patients is still unknown.

ELIGIBILITY:
Inclusion Criteria:

Generally healthy children aged between 3-5 years with no remarkable medical history.

Exclusion Criteria:

1. Children with the presence of caries of ICDAS code 3, 4, 5, or 6 on other primary teeth.
2. Children who had received professional fluoride application in the past 6 months.
3. Children with serious systemic disease or taking long term medication.
4. Children who are uncooperative or refuse the treatment.
5. Second primary molars that are (i) with caries in dentin indicated by ICDAS code 4, 5 or 6; (ii) partially erupted; (iii) with fillings and/or sealants; and (iv) hypoplastic or hypomineralized.

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 348 (Estimated)
Dates: Start 2018-04-11 (Actual); Primary Completion 2021-08-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Caries increment | 24 months
  Carious cavity development into dentin (ICDAS code 4, 5 and 6) on the occlusal surfaces of primary second molars over time.

SECONDARY OUTCOMES:
Sealant retention | 24 months
  Retention of GIS on included primary second molar

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Kar Yung Yiu, FHKAM,FCDSHK, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ahovuo-Saloranta A, Hiiri A, Nordblad A, Worthington H, Makela M. Pit and fissure sealants for preventing dental decay in the permanent teeth of children and adolescents. Cochrane Database Syst Rev. 2004;(3):CD001830. doi: 10.1002/14651858.CD001830.pub2. PMID 15266455
- [Background] American Academy of Pediatric Dentistry. Guideline on caries-risk assessment and management for infants, children, and adolescents. Pediatr Dent. 2013 Sep-Oct;35(5):E157-64. No abstract available. PMID 24290544
- [Background] Marinho VC. Cochrane reviews of randomized trials of fluoride therapies for preventing dental caries. Eur Arch Paediatr Dent. 2009 Sep;10(3):183-91. doi: 10.1007/BF03262681. PMID 19772849
- [Background] Ahovuo-Saloranta A, Forss H, Hiiri A, Nordblad A, Makela M. Pit and fissure sealants versus fluoride varnishes for preventing dental decay in the permanent teeth of children and adolescents. Cochrane Database Syst Rev. 2016 Jan 18;2016(1):CD003067. doi: 10.1002/14651858.CD003067.pub4. PMID 26780162
- [Derived] Ying Lam PP, Sardana D, Luo W, Ekambaram M, Man Lee GH, Man Lo EC, Yung Yiu CK. Glass Ionomer Sealant versus Fluoride Varnish Application to Prevent Occlusal Caries in Primary Second Molars among Preschool Children: A Randomized Controlled Trial. Caries Res. 2021;55(4):322-332. doi: 10.1159/000517390. Epub 2021 Jul 20. PMID 34284374

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-17): https://cdn.clinicaltrials.gov/large-docs/54/NCT04163354/Prot_SAP_000.pdf